CLINICAL TRIAL: NCT07343219
Title: Effects of Root Extract Ashwagandha (KSM-66) on Physiological Stress, Perception of Recovery and Muscle Strength in Youth Elite Footballers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sports Performance and Applied Research in Trials and Analysis (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20251103
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Performance; Recovery; Strength; Aerobic Endurance
Keywords: ashwagandha; football; strength; recovery
MeSH Terms: interventions — Starch

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind and placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwagandha root extract (Experimental): 450 mg Ashwagandha root extract
  Interventions: Dietary Supplement: Root extract Ashwagandha
- Placebo (Placebo Comparator): 450 mg corn starch
  Interventions: Other: Corn Starch

INTERVENTIONS:
Dietary Supplement: Root extract Ashwagandha — 450 mg Ashwagandha root extract
  Arms: Ashwagandha root extract
Other: Corn Starch — 450 mg corn starch
  Arms: Placebo

SUMMARY:
This trial examines if six weeks of taking 450 mg Ashwagandha root extract affects exercise performance and recovery in youth male elite football players.

Ashwagandha root extract is increasingly used by athletes, but controlled research in adolescent athletes is limited and the majority of evidence is in an adult population. This study will assess short-term responses in youth players.

Participants will be randomly assigned to take either Ashwagandha root extract or a placebo once daily for six weeks. Players will complete training-based tests, provide saliva samples and complete a short, validated questionnaire on perception of wellness. Any adverse events will be documented and reported.

DETAILED DESCRIPTION:
The objective of this trial is to learn whether a short period of taking 450mg of Ashwagandha root extract affects performance, recovery, muscle strength and wellbeing in youth male elite football players.

The researchers are studying Ashwagandha root extract as it is increasingly used by athletes and the general population of varying ages for well-being, performance and recovery purposes, despite a lack of controlled research examining its effects in adolescent athletes. Most existing evidence comes from adult populations, and it remains unclear whether similar physiological and perceptual responses occur in adolescents engaged in structured training.

The main questions the study aims to answer are:

Does taking Ashwagandha root extract change stress levels measured through saliva in youth elite footballers?

Does it affect muscle strength, recovery, sleep, or muscle soreness?

Participants will be randomly assigned to take either Ashwagandha root extract or a placebo once a day for six weeks. During the study, players will complete strength and fitness tests during usual training time, then provide saliva samples afterwards. Short questionnaires will be solicited the day after about how they feel. Any adverse events that occur during the study will be documented and reported.

ELIGIBILITY:
Inclusion Criteria:

* Male youth football player
* Classified as 'healthy' and 'free of disease'
* Actively training with the selected football academy

Exclusion Criteria:

* Lack of signed consent form
* No active use of medication
* No active use of ergogenic aids
* Allergies to nightshades

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Change in Salivary Cortisol Concentration from Baseline to 6 Weeks | 6 weeks

SECONDARY OUTCOMES:
Change in Salivary Alpha Amylase from Baseline to 6 Weeks | 6 weeks
Change in Handgrip Strength (kg) from Baseline to 6 Weeks | 6 weeks
  Hand grip strength using CAMRY dynamometer
Change in Countermovement Jump Height (cm) from Baseline to 6 Weeks | 6 weeks
Change in 1 km Time Trial Completion Time (seconds) from Baseline to 6 Weeks | 6 weeks
  Maximal effort run of 1km
Perception of sleep quality | Baseline to 6 weeks
  Sleep quality will be assessed using the sleep domain of the Hooper Index, which is one of four domains within the questionnaire (fatigue, stress, delayed onset muscle soreness, and sleep). The sleep item is rated on a 10-point scale (1 to 10), where 1 indicates very, very good sleep and 10 indicates very, very poor sleep. This domain will be analysed independently as a subset of the Hooper Index, rather than as part of the total score.
Perception of stress | Baseline to 6 weeks
  Perceived stress will be assessed using the sleep domain of the Hooper Index, which is one of four domains within the questionnaire (fatigue, stress, delayed onset muscle soreness and sleep). The stress item is rated on a 10-point scale (1 to 10), where 1 indicates very, very good and 10 indicates very, very poor. This domain will be analysed independently as a subset of the Hooper Index, rather than as part of the total score.
Perception of muscle soreness | Baseline to 6 weeks
  Perceived muscle soreness will be assessed using the sleep domain of the Hooper Index, which is one of four domains within the questionnaire (fatigue, stress, delayed onset muscle soreness and sleep). The muscle soreness item is rated on a 10-point scale (1 to 10), where 1 indicates very, very good and 10 indicates very, very poor. This domain will be analysed independently as a subset of the Hooper Index, rather than as part of the total score.
Perception of fatigue | Baseline to 6 weeks
  Perceived fatigue will be assessed using the sleep domain of the Hooper Index, which is one of four domains within the questionnaire (fatigue, stress, delayed onset muscle soreness and sleep). The fatigue item is rated on a 10-point scale (1 to 10), where 1 indicates very, very good and 10 indicates very, very poor. This domain will be analysed independently as a subset of the Hooper Index, rather than as part of the total score.
Overall Hooper Index Score | Baseline to 6 weeks
  Perceived recovery will be assessed using the Hooper Index, which evaluates four domains: fatigue, stress, delayed onset muscle soreness (DOMS) and sleep quality. Each domain is rated on a 10-point scale (1 to 10), where 1 indicates very, very good and 10 indicates very, very poor. The total Hooper Index score is calculated by summing the four domains, resulting in a possible range of 4 to 40, with higher scores indicating worse perceived recovery, greater fatigue and stress, and lower scores indicating better recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia C Coope, PhD, Study Director — Blanquerna Institute
Locations (1):
- Fulham Football Club, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to primary and secondary outcomes will be shared with other sports nutrition researchers upon reasonable request. Data sharing will be subject to ethical approval, data protection requirements, and safeguarding considerations, and will exclude any information that could identify participants.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bonilla DA, Moreno Y, Gho C, Petro JL, Odriozola-Martinez A, Kreider RB. Effects of Ashwagandha (Withania somnifera) on Physical Performance: Systematic Review and Bayesian Meta-Analysis. J Funct Morphol Kinesiol. 2021 Feb 11;6(1):20. doi: 10.3390/jfmk6010020. PMID 33670194
- [Background] Mishra RK, Trivedi R, Pandya MA. A clinical study of Ashwagandha ghrita and Ashwagandha granules for its Brumhana and Balya effect. Ayu. 2010 Jul;31(3):355-60. doi: 10.4103/0974-8520.77164. PMID 22131739
- [Background] Petroczi A, Naughton DP, Pearce G, Bailey R, Bloodworth A, McNamee M. Nutritional supplement use by elite young UK athletes: fallacies of advice regarding efficacy. J Int Soc Sports Nutr. 2008 Dec 15;5:22. doi: 10.1186/1550-2783-5-22. PMID 19077317